CLINICAL TRIAL: NCT03725319
Title: Retrospective Study on Treatment of Post Sphincterotomy-bleeding by Epinephrine-injection Versus Insertion of an Endoprosthesis: a Single Center Experience Over 16 Years With 5698 ERCPs
Brief Title: Treatment of Post Sphincterotomy-bleeding by Epinephrine-injection Versus Insertion of an Plastic Stent
Status: Completed | Type: Observational
Sponsor: Theresienkrankenhaus und St. Hedwig-Klinik GmbH (Other)
Responsible Party: Principal Investigator, Daniel Schmitz, Assistant medical director, Theresienkrankenhaus und St. Hedwig-Klinik GmbH
Other Study IDs: PSB Epiverstent 01
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Endoscopic Biliary Sphincterotomy; Bleeding
Keywords: Endoscopic Biliary Sphincterotomy; Endoscopic Retrograde Cholangiopancreatography; Bleeding; Epinephrine; Stent
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epinephrin injection: Diluted Epinephrin (1:100) in small amounts from 1 to 5 ml is injected into apex of the papilla to stop post sphincterotomy-bleeding
- Plastic stent insertion: A plastic stent (diameter: 8-11,5F and length of 50 -100mm) is inserted into the common bile duct to stop post sphincterotomy-bleeding

SUMMARY:
Post sphinterotomy-bleeding (PSB) occurs in 1-2 % of Endosocpic Retrograde Cholangiopancreaticography (ERCP) and usually needs no blood transfusion after endoscopic therapy but can be life-threatening in some rare cases.

There are no prospective comparative studies concerning the endoscopic treatment of PSB due to the rarity of the incident.

Insertion of an endoprosthesis in the common bile duct may be more effective than Epinephrin-injection into the papilla which is the therapy of first choice.

A retrospective single centre analysis on both used methods over a study period of 16 years shall be performed.

DETAILED DESCRIPTION:
Post sphinterotomy-bleeding (PSB) occurs in 1-2 % of Endosocpic Retrograde Cholangiopancreaticography (ERCP) and usually needs no blood transfusion after endoscopic therapy but can be life-threatening in some rare cases.

The increasing use of antiplatelet and/or anticoagulant therapies enhances the risk of PSB.

There are no prospective comparative studies concerning the endoscopic treatment of PSB due to the rarity of the incident.

Insertion of an endoprosthesis in the common bile duct may be more effective than Epinephrin-injection into the papilla which is the therapy of first choice.

A retrospective single centre analysis on both used methods over a study period of 16 years shall be performed.

In detail, clinical success and safety of the procedure, re-bleeding rate, number of re-interventions and days of hospital stay will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Post sphincterotomy bleeding (PSB) of the papilla (time frame: from procedure up to ten days after the procedure)
* Treatment of PSB by epinephrine-injection or insertion of a plastic stent into the common bile duct

Exclusion Criteria:

* Pregnant and/or lactating women
* Complete patient record is not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All documented ERCPs in the single centre institution database are systematically screened for post sphincterotomy-bleeding in the time period from 1.1.2002 to 29.10.2018
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Clinical success | From the successful endocopic treatment of post sphincterotomy-bleeding up to 30 days in the follow up
  No re-bleeding occurs in the follow-up that requirers a further interventional treatment of re-bleeding (any endoscopic, radiological embolization or surgery): yes/no
Re-interventions | From the endoscopic treatment of post-sphincterotomy-bleeding up to three months
  Amount of endoscopic re-interventions (further endoscopic therapy of re-bleeding of the papilla, removal or exchange of the plastic stent): number (n)
Hospital stay after treatment | From the endoscopic treatment of post-sphincterotomy-bleeding up to 30 days
  Hospital stay (days) after treatment of post sphincterotomy-bleeding

SECONDARY OUTCOMES:
Post ERCP-pancreatitis | From the endoscopic treatment of post-sphincterotomy-bleeding up to three days
  Any kind of post ERCP-pancreatitis that occurs after treatment of post sphincterotomy-bleeding and can be refered to this treatment (patients with cannulated pancreatic duct are excluded): yes/no
Increasing of cholestasis parameters | From treatment of post-sphincterotomy-bleeding up to three days
  Any kind of cholestasis measured by an increase of bilirubin level (mg/dl) after the treatment of post-sphincterotomy-bleeding that can be refered to this treatment (patients with unsuccesful endoscopic drainage/stone extraction are excluded): yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Schmitz, Dr.med., Principal Investigator — Theresienkrankenhaus und St.Hedwigsklinik GmbH, Bassermannstr.1, 68165 Mannheim
Locations (1):
- Tertiary referral hospital: Theresienkrankenhaus und St. Hedwig Hospital, Academic, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andriulli A, Loperfido S, Napolitano G, Niro G, Valvano MR, Spirito F, Pilotto A, Forlano R. Incidence rates of post-ERCP complications: a systematic survey of prospective studies. Am J Gastroenterol. 2007 Aug;102(8):1781-8. doi: 10.1111/j.1572-0241.2007.01279.x. Epub 2007 May 17. PMID 17509029
- [Background] Freeman ML, Nelson DB, Sherman S, Haber GB, Herman ME, Dorsher PJ, Moore JP, Fennerty MB, Ryan ME, Shaw MJ, Lande JD, Pheley AM. Complications of endoscopic biliary sphincterotomy. N Engl J Med. 1996 Sep 26;335(13):909-18. doi: 10.1056/NEJM199609263351301. PMID 8782497
- [Background] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Background] Matsushita M, Hajiro K, Takakuwa H, Nishio A. Effective hemostatic injection above the bleeding site for uncontrolled bleeding after endoscopic sphincterotomy. Gastrointest Endosc. 2000 Feb;51(2):221-3. doi: 10.1016/s0016-5107(00)70425-1. No abstract available. PMID 10650275